CLINICAL TRIAL: NCT00454415
Title: Prospective Study of Dietary Factors, BMI, and Risk of Asthma in Children
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Carlos A. Camargo, Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 1376; R01HL084401-01A1 (NIH)
Record Dates: First submitted 2007-03-28; First posted 2007-03-30 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Asthma
Keywords: Diet; Body Mass Index; BMI
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Asthma is a common illness among children in the United States. While there are many known causes of asthma, including tobacco smoke, pollen, dust, or other allergens, the exact cause of asthma in some individuals remains unknown. This study will examine the role that specific dietary factors and body mass index (BMI) play in the development of childhood asthma.

DETAILED DESCRIPTION:
Asthma prevalence has steadily increased in the United States since the early 1980s, but the exact cause of this increase remains unknown. It is estimated that at least 8% of Americans have asthma. Although anti-inflammatory medications have proven effective for decreasing asthma exacerbations, there are few treatment options available to prevent the initial onset of the disease. Dietary factors and BMI may play a role in the development of asthma. Specifically, individuals who eat foods containing antioxidants (e.g., vitamin C, vitamin E, and carotenoids), n-3 polyunsaturated fatty acids (e.g., fish oils), and vitamin D may have a decreased risk of developing asthma, while individuals with higher BMI ratios may have an increased asthma risk. The purpose of this study is to evaluate the relationship among dietary factors, BMI, and the incidence of asthma among children.

This study will enroll children participating in the Growing Up Today study and children of nurses who are participating in the Nurses Health Study II. Researchers will analyze participants' previously completed questionnaires on dietary intake, physical activity, height, weight, and the presence of physician-diagnosed asthma. All participants with physician-diagnosed asthma will receive an additional asthma questionnaire. A small portion of these participants will also have their medical records reviewed by study researchers, and mothers of these children will be asked to complete a questionnaire. Additionally, a questionnaire will be sent to and completed by children who do not have asthma and their mothers.

ELIGIBILITY:
Inclusion Criteria:

* Children of women in the Nurses Health Study II (NHS2)
* Participated in the Growing Up Today study

Exclusion Criteria:

* None

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: U.S. children
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
incident asthma | childhood

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A. Camargo, MD, DrPH, Principal Investigator — Channing Laboratory, Brigham and Women's Hospital
Locations (1):
- Channing Laboratory, Brigham and Women's Hospital, Boston, Massachusetts, United States